CLINICAL TRIAL: NCT00714376
Title: Phase II Single Center Study of Docetaxel for Clinically Asymptomatic High Risk Prostate Cancer Patients With an Early Rising PSA Following Radical Prostatectomy
Brief Title: Phase II Study of Docetaxel for Clinically Asymptomatic High Risk Prostate Cancer Patients
Acronym: TAX1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Prematurely terminated due to financial considerations
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Yves Fradet, Urologist-Oncologist, CHU de Quebec-Universite Laval
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Project 5.2.08.02
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; High-risk prostate cancer; Radical prostatectomy; Early rising PSA; Taxotere; Docetaxel
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel (Experimental): Docetaxel (Taxotere) 75 mg/m² IV every 3 weeks for 8 cycles.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m2 iv every 3 weeks for 8 cycles
  Other Names: Taxotere

SUMMARY:
The purpose of this study is to assess the response to Taxotere (docetaxel) chemotherapy given as a primary treatment to patients with early and rapid PSA rising after prostatectomy for high risk disease.

DETAILED DESCRIPTION:
Patients with high-risk prostate cancer have a high probability of PSA failure after radical prostatectomy. However, more than half of these patients will remain free of PSA recurrence for more than 10 years. To the contrary, patients with early PSA recurrence and a doubling time less than 10 months have a mortality rate approaching 50% at 10 years despite hormone therapy. Although androgen deprivation therapy (ADT) remains the standard treatment for patients with early and rapidly rising PSA after prostatectomy, this treatment is not curative on the long term for most patients. The recent demonstration of activity of Taxotere (docetaxel) in a high proportion of patients with advanced metastatic disease has stimulated a great interest in it use at an earlier stage of the disease. Recent studies performed in animal models of prostate cancer suggested that the response rate of prostate cancer cells to docetaxel-induced cell death was significantly enhanced by androgen stimulation in AR-positive, androgen-dependent prostate cancer cells (i.e. before ADT). Therefore, this protocol proposes to assess the response rate to primary Taxotere chemotherapy in patients with early and rapid PSA rising after prostatectomy for high risk disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of prostate adenocarcinoma on a radical prostatectomy.
2. Prior radical prostatectomy within less than 2 years from the time of first PSA rise.
3. Demonstration of biochemical recurrence based on a PSA detectable >0.03 less than 24 months after radical prostatectomy and confirmed on 2 additional tests.
4. PSA doubling time over three values must be <= 9 months for PSA >=0.4 and PSA <=10. If PSA is >10, there is no need for PSA doubling time.
5. Karnofsky performance status (KPS) >=70%
6. Adequate organ function as defined by hemogram with haemoglobin >8.0, platelet >100 000, white blood cell >3,500, creatinine clearance >=60 cc/min and normal liver function tests.
7. Neoadjuvant hormone therapy prior to radical prostatectomy is allowed provided that the total duration of therapy did not exceed 6 months.
8. Subjects must have signed an informed consent document stating that they understand the investigational or nature of the proposed treatment.
9. Subjects must be willing and able to comply with scheduled visits, treatment plans, laboratory tests and other procedures.

Exclusion Criteria:

1. Clinical significant cardiac disease (New York Heart Association Class III/IV), or severe debilitating pulmonary disease.
2. Uncontrolled serious active infection.
3. Anticipated duration of life less than 2 years.
4. Less than 5-year history of successful treatment for other cancers or concurrent active non prostate cancer other than non melanoma dermatologic tumors and non-muscle invasive bladder tumors.
5. Peripheral neuropathy >=2 grade 2
6. Concurrent experimental treatment or involvement in other clinical trials involving drugs.
7. Other severe acute or chronic medical conditions including psychiatric diseases or significant laboratory abnormality requiring further investigation that may cause undue risk for the subject's safety.
8. Subjects who participated in another clinical study/received investigational product within 30 days of screening for this study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the rate of partial and complete biochemical response to 8 cycles of Taxotere in patients with early (<2 years) PSA recurrence after radical prostatectomy with a PSA doubling time of <=9 months. | 3 to 6 months

SECONDARY OUTCOMES:
To evaluate the response rate to subsequent androgen deprivation therapy in patients not responding and in those having a biochemical recurrence after complete response. | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yves Fradet, MD, Principal Investigator — Centre Hospitalier Universitaire de Quebec (CHUQ); Pierre Ouellet, MD, Principal Investigator — CHU de Quebec-Universite Laval
Locations (1):
- Centre de recherche clinique et evaluative en oncologie, L'Hôtel-Dieu de Québec-CHUQ, Québec, Quebec, Canada